CLINICAL TRIAL: NCT03053557
Title: Social Skills Coach: An Innovative Multi-Platform Device to Address Social Impairments
Brief Title: Testing a New Device to Advance the Use of Social Skills Training With Mental Health Consumers and Clinicians
Acronym: SST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Social Innovation, Massachusetts (Other)
Collaborators: University of Maryland (Other); VA Maryland Health Care System (U.S. Federal Agency); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Social Skills Coach; 1R43MH113424-01 (NIH)
Record Dates: First submitted 2017-02-09; First posted 2017-02-15 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Schizophrenia Spectrum and Other Psychotic Disorders
Keywords: mental health consumers
MeSH Terms: conditions — Schizophrenia Spectrum and Other Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: Convergent parallel mixed methods
Who Masked: Outcomes Assessor
Masking Description: Research assistants who conduct assessments with participants will be blinded as to whether participants have been assigned to the intervention or control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social Skills Coach (Experimental): The Social Skills Coach arm of the study will be provided access, instruction, and support for using the newly developed multi-platform device to address social impairments among individuals with schizophrenia, based on the evidence-based Social Skills Training (SST) intervention.
  Interventions: Behavioral: Social Skills Coach
- Social Skills Training course (No Intervention): Social Skills Training classes are widely available and regularly used in the study setting. As such, this group will serve as a treatment as usual control group.

INTERVENTIONS:
Behavioral: Social Skills Coach — Social Skills Coach is a multi-platform interactive device that engages users with information and skills learned in social skills training programs. The program includes a web application and provider dashboard and encourages users to practice skills on the app and use them in the real world and then report how the application of skills was experienced.
  Arms: Social Skills Coach

SUMMARY:
This study aims to test a new device called the Social Skills Coach that is being created to help mental health consumers with social skills and community functioning. People diagnosed with schizophrenia and clinicians will be included as participants in this study. Mental health consumers (diagnosed with schizophrenia) will be randomly assigned to either test the new device or to participate in a social skills training course. Data will be collected from participants through surveys before participants either use the device or participate the course and afterwards. Individual interviews will be conducted with a sub sample of mental health consumers and clinicians. The study looks to test the credibility and acceptability of the new device to help mental health consumers and clinicians. it will also influence future research.

DETAILED DESCRIPTION:
This phase I pilot study tests the feasibility, credibility, and acceptability of the prototype version of Social Skills Coach in terms of its use among mental health consumers and clinicians. The intervention aims to improve social and daily living skills and community functioning among people diagnosed with schizophrenia spectrum disorder. A mixed methods approach will be taken to collect quantitative data at baseline and follow-up. Quantitative data collection includes the use of surveys that comprise validated instruments. Qualitative data collection will occur at the end of the study and will include the use of semi-structured interviews to capture experiential information. Study participants will be randomly assigned to either a social skills training course (control group) or to a study arm using the Social Skills Coach program (treatment group). The study aims to demonstrate proof of concept for a larger effectiveness trial.

ELIGIBILITY:
Inclusion Criteria:

* Chart diagnosis of schizophrenia spectrum disorder, ability to provide consent, and independent living in the community.
* We will obtain written informed consent, and the consent procedure will include an evaluation of capacity to provide consent

Exclusion Criteria:

* Under age 21 or not able to provide consent.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Feasibility: 90% recruitment, 75% data completed, 80% technical problems solved | 4 weeks post intervention
  Study Process: Recruitment, Retention, Troubleshooting
Credibility: Mean greater than 6 on Expectancy Rating Scale | 4 weeks post intervention
  Expectancy Rating Scale collected from client participants
Acceptability: 80% of participants engage at least once; 50% of group attendees enter personalized goals; 50% of participants enter an evaluation goal | 4 weeks post intervention
  Web diagnostics and through Qualitative interviews with client participants and SST trainer participants

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Olivet, MA, Principal Investigator — Center for Social Innovation
Locations (1):
- Center for Social Innovation, Needham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Data will be password protected and stored on secure severs. Access will be restricted to only the study team. When data is shared between team members it will be deidentified. All researchers on this project will have completed human subjects training and training specific to study protocols.